CLINICAL TRIAL: NCT02290132
Title: Hematology , Shanghai Jiaotong University Affiliated Shanghai First People's Hospital, Shanghai, China
Brief Title: ATG Could Improve the Outcome Of Hematopoietic Stem Cell Transplant in Patients With Highly Aggressive T Cell Tumors
Acronym: HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Tang-Du Hospital (Other); The First Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yang Jun, hematology , Shanghai Jiaotong University affiliated Shanghai First People's Hospital, shanghai, China, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 2013（56）
Record Dates: First submitted 2014-10-13; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: acute lymphoblastic leukemia; lymphoblastic lymphoma; stem-cell transplant; T-cell lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell | interventions — thymoglobulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- highly aggressive T cell tumors: The study is to research the outcome of Rabbit Anti-human Thymocyte Globulin (ATG)based myeloablative conditioning regimen after allo-HSCT in patients with highly aggressive T-cell tumors.
  Interventions: Drug: Rabbit Anti-human Thymocyte Globulin (ATG)

INTERVENTIONS:
Drug: Rabbit Anti-human Thymocyte Globulin (ATG) — The conditioning regimen in this study consisted of Rabbit antithymocyte globulin (ATG 2.5 mg/kg×4 days) , total-body irradiation (10 Gy in five fractions), cyclophosphamide (60 mg/kg×2 days) and etoposide or teniposide (30-40mg/kg) .
  Other Names: r-ATG

SUMMARY:
The clinical application and effect of ATG based myeloablative conditioning regimen after allogeneic hematopoietic stem cell transplantation in adult patients with aggressive T-cell lymphomas.

DETAILED DESCRIPTION:
Aggressive T-cell lymphomas (ATCLs), including peripheral T-cell lymphoma and T lymphoblastoid cell lymphoma/leukemia, represent 10% to 15% of non-Hodgkin's lymphomas (NHLs) in adults(1). ATCLs show a worse prognosis than that of B-cell lymphomas. Myeloablative allogeneic stem cell transplantation (allo-SCT) may be the only way to cure these patients, but the recurrence of the primary disease after transplantation is still an important prognostic factor (2). Optimizing the conditioning regimen is always the research hot topics in hematology fields. Polyclonal anti-thymocyte globulin (rabbit anti-thymocyte globulin, r-ATG) are currently used to prevent graft-versus -host(GVHD) disease in allogeneic stem cell transplantation, and also widely used for the prevention and treatment of acute rejection after solid organ transplant because of its strong immunomodulatory effects. ATG is used in allogeneic SCT for the prophylaxis of graft versus host disease by in vivo T cell depletion, including the complement-dependent cytotoxic response, antibody-dependent cell-mediated cytotoxicity, the opsonophagocytic role of phagocytic cells and induced apoptosis(3). But some scholars reported the ATG delayed immune reconstitution and hematologic reconstitution and leaded to the increase of the incidence of virus and fungal infections after transplantation. But it is often curable and does not affect the overall survival and quality of life of the patients (4). Because of its strong immune suppression and regulation, also on the basis of the above facts, ATG as GVHD prophylaxis is generally limited to the unrelated donor, or human leukocyte antigen（HLA）-mismatched related donor transplantation. But There are many issues still need to be studied. ATG has shown efficacy in preventing acute GVHD（aGVHD) in allo-SCT, but its efficacy in chronic GVHD (cGVHD) and long-term outcomes remains controversial. A systematic review and meta-analysis from Du k et al（5） reported that prophylactic use of ATG exerted a favorable effect in reducing cGVHD without survival impairment in a long term, although a higher relapse rate is a major threat.

Does the ATG also have the killing effect on the tumor cells of the lymphatic system? The vitro studies have confirmed this point recently. Grüllich(6) et al and the investigators study(7) both found that ATG can inhibit the proliferation and induce high level of apoptosis in the human lymphoblastic cell lines, such as Jurkat, Daudi, DG-75 , and myeloblastic cell lines K562, HL-60, KG1, and U937. ATG also has pro-apoptotic activity against the majority of primary leukemia cells, particularly those cells from lymphatic origin. In addition, ATG will not result in apoptosis of normal hematopoietic cells. Low-dose ATG can also stimulate normal hematopoietic colony growth. Therefore, ATG may be used as anti-lymphocyte tumor bio-therapeutics (such as rituximab) to increase the role of chemo-radiotherapy in the conditioning regimen. And ATG can remove the residual tumor lesions, which reduced the rate of tumor recurrence after transplantation. Although the vitro studies have clarified the role of ATG on the tumor cells of the lymphatic system, but no relevant reports on the anti-tumor effect of ATG in allo-SCT have been published. Further clinical observation need to be conducted.

As noted earlier, a higher relapse rate may be a major threat after ATG use（5）.In China, the conventional dose of 2.5mg/kg/day, 2-3 days of Thymoglobulin is commonly used as GVHD prophylaxis in the unrelated donor, or HLA-mismatched related donor transplantation but not in the HLA matched related donor transplantation (8). In order to observe the anti-tumor effect of this conditioning regimen in the aggressive T-cell lymphomas patients(including peripheral T-cell lymphoma and T lymphoblastoid cell lymphoma/leukemia, complete remission, partial remission, relapse after remission or refractory recurrent invasive patients), the investigators improved the drugs of conditioning regimen and increased the Thymoglobulin dose in the conditioning regimen for four days 10mg/kg total even in the HLA matched related donor transplantation. The purpose of this clinical trial is to reduce the incidence of GVHD at the same time does not increase the recurrence of the primary disease. The investigators expect that this ATG based conditioning regimen does play anti-tumor effect, reduce primary disease recurrence after transplantation, improve disease-free survival (DFS) and overall survival rate (OS) , as well as reduce the incidence and severity of GVHD, but the incidence of infection need to be observed.

ELIGIBILITY:
Inclusion Criteria:

* According to the World Health Organization (WHO) classification, diagnosis of T cell tumor of lymphatic system sources (including peripheral T-cell lymphoma and T lymphoblastoid cell lymphoma/leukemia) confirmed by pathological examination, morphology, cytochemistry, immunophenotyping and chromosome examination, molecular biology including complete remission, partial remission, relapse after remission or refractory recurrent invasive patients
* 18 to 60 years old. Male or female
* Performance status scores no more than 2 (ECOG criteria).
* Adequate organ function as defined by the following criteria:

alanine transaminase （ALT）, aspartate transaminase（AST） and total serum bilirubin <2×ULN (upper limit of normal)

* Serum creatinine and blood urea nitrogen(BUN) <1.25×ULN.
* Adequate cardiac function without acute myocardial infarction, arrhythmia or atrioventricular block, heart failure, active rheumatic heart disease and cardiac dilatation(the patients has been improved after treatment of the disease and are not expected to affect transplant can include in the study).
* Absence of any other contraindications of stem cell transplantation.
* Willingness and ability to perform HSCT.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Presence of any condition inappropriate for HSCT.
* Life expectancy < 3 months because of other severe diseases.
* Presence of any fatal disease, including respiratory failure, heart failure, liver or kidney function failure et al.
* Uncontrolled infection.
* Pregnancy or breastfeeding. 6．Has enrolled in anther clinical trials 7．Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: According to the World Health Organization (WHO) classification,study population is diagnosis of T cell tumor of lymphatic system sources (including peripheral T-cell lymphoma and T lymphoblastoid cell lymphoma/leukemia) confirmed by pathological examination, morphology, cytochemistry, immunophenotyping and chromosome examination, molecular biology including complete remission, partial remission, relapse after remission or refractory recurrent invasive patients
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Progress free surviva(PFS) rate at 2 years | 2 YEARS
  PFS were defined as the time from stem-cell infusion to relapse, disease progression,or death from any cause

SECONDARY OUTCOMES:
Leukocyte engraftment | 1 MONTH
  Leukocyte engraftment:(was defined as the first of three consecutive days of peripheral white blood count >1000/ul.
Platelet engraftment | 1 MONTH
  Platelet engraftment:(was defined as the first of seven consecutive days of platelet counts of >50000/ul.
Donor chimerism: | 2 YEARS
  Quantitative chimerism analyzes were performed using short-tandem-repeat-based polymerase chain reaction technique sat regular intervals for every 4 weeks after allografting in bone marrow.
Relapse incidence (RI) | 2 YEARS
  1. T lymphoblastoid cell lymphoma/leukemia: Bone marrow blasts > 20% 2.peripheral T-cell lymphoma: any increased >50% in the sum of the diameter of any measurable lesions or the appearance of a new lesion.）
Overall survival rate | 2 YEARS
  OS were defined as the time from stem-cell infusion to death from any cause)
Transplant related mortality(TRM) | 2 YEARS
  TRM were defined as death within 100 days of high-dose therapy not related to the disease,relapse or progression

CONTACTS AND LOCATIONS:
Overall Officials: liu guohua, doctor, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's HOSPITAL, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Rudiger T, Weisenburger DD, Anderson JR, Armitage JO, Diebold J, MacLennan KA, Nathwani BN, Ullrich F, Muller-Hermelink HK; Non-Hodgkin's Lymphoma Classification Project. Peripheral T-cell lymphoma (excluding anaplastic large-cell lymphoma): results from the Non-Hodgkin's Lymphoma Classification Project. Ann Oncol. 2002 Jan;13(1):140-9. doi: 10.1093/annonc/mdf033. PMID 11863096
- [Background] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005
- [Background] Mohty M. Mechanisms of action of antithymocyte globulin: T-cell depletion and beyond. Leukemia. 2007 Jul;21(7):1387-94. doi: 10.1038/sj.leu.2404683. Epub 2007 Apr 5. PMID 17410187
- [Background] Du K, Hu Y, Wu K, Huang H. Long-term outcomes of antithymocyte globulin in patients with hematological malignancies undergoing myeloablative allogeneic hematopoietic cell transplantation: a systematic review and meta-analysis. Clin Transplant. 2013 Mar-Apr;27(2):E91-E100. doi: 10.1111/ctr.12091. Epub 2013 Feb 6. PMID 23383989
- [Background] Grullich C, Ziegler C, Finke J. Rabbit anti T-lymphocyte globulin induces apoptosis in peripheral blood mononuclear cell compartments and leukemia cells, while hematopoetic stem cells are apoptosis resistant. Biol Blood Marrow Transplant. 2009 Feb;15(2):173-82. doi: 10.1016/j.bbmt.2008.11.014. PMID 19167677
- [Background] Meijer E, Cornelissen JJ, Lowenberg B, Verdonck LF. Antithymocyteglobulin as prophylaxis of graft failure and graft-versus-host disease in recipients of partially T-cell-depleted grafts from matched unrelated donors: a dose-finding study. Exp Hematol. 2003 Nov;31(11):1026-30. doi: 10.1016/s0301-472x(03)00204-2. PMID 14585365
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Result] Liu H, Qin Y, Wang X, Xie K, Yang Y, Zhu J, Zhao C, Wang C. Polyclonal rabbit antithymocyte globulin induces apoptosis and has cytotoxic effects on human leukemic cells. Clin Lymphoma Myeloma Leuk. 2012 Oct;12(5):345-54. doi: 10.1016/j.clml.2012.05.006. Epub 2012 Jun 6. PMID 22677206